CLINICAL TRIAL: NCT03484910
Title: Application of Biofeedback Combined With Cycling Exercise in the Patients With Osteoarthritis of the Knee
Brief Title: Biofeedback With Cycling Exercise in OA Knee Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hsiu-Chen Lin, Associate Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMUH106-REC3-001
Record Dates: First submitted 2018-03-19; First posted 2018-04-02 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Exercise Therapy; Osteoarthritis Of Knee; Biofeedback
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BFB group (Experimental): Exercise therapy - Six-week training program of stationary cycling with a real-time visual EMG biofeedback
  Interventions: Other: Exercise therapy
- CON group (Active Comparator): Exercise therapy - Six-week training program of stationary cycling without EMG biofeedback
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Exercise therapy — Six-week training program of stationary cycling with / without a real-time visual EMG biofeedback

SUMMARY:
Osteoarthritis (OA) is one of the most common joint diseases causing pain, muscle weakness and disability in older population. Quadriceps muscle weakness is one of the recognized risk factors for the development and the progression of the disease. Increasing the muscle strength could actually bring many benefits to the knee OA patients. The purposes of this study are 1) to investigate the effects of combining the EMG biofeedback technique into a stationary cycling exercise on the activities of vastus medialis (VM) in people with medial compartment knee OA; 2) To investigate the efficiency of a 6-week cycling exercise program on improving of quadriceps muscle strength and endurance, physical functions and pain in these patients and compare between the conditions of with or without EMG biofeedback; 3) To determine the relationships between the muscle activities and the kinematics of the knee joint during this cycling exercise program; and therefore to find the mechanism of the improvement on muscle activities in the intervention of cycling combining EMG biofeedback. In this study, we will enroll the knee OA patients from our hospital, and they will be randomly assigned either to the control group, who will cycle without biofeedback, or the biofeedback group, who will cycle with a real-time visual EMG biofeedback, during the six-week training program. The exercise program consisted of a 5-minute warm-up with low-resistance cycling, 30-minute moderate-resistance cycling exercise, and 5-minute cool down session. . The knee adduction angle, quadriceps strength and endurance, KOOS Chinese version, VAS scale will also be measured at baseline and after six weeks of intervention. Mixed-model repeated measure analysis of variance (ANOVA) will be used to determine if there are any differences in the kinematic, myoelectric, muscle strength and endurance. It is hoped that the results of this study could provide information regarding the proper and efficient training strategy for the OA knee patients, and deliver the concepts of proper exercise technique to enhance health in the community.

ELIGIBILITY:
Inclusion Criteria:

* the OA knee patients are those who had medial compartment tibiofemoral osteoarthritis in either one or both of their knees, had at least a grade 2 on the Kellgren-Lawrence score, which was verified with radiographs and a diagnosis by a physician

Exclusion Criteria:

* if the participant had been diagnosed with OA in the hip or ankle joints, had a lower extremity joint replacement, had knee joint arthroscopic surgery or intra-articular injections within 3 months prior to testing, had systemic inflammatory arthritis such as rheumatoid or psoriatic arthritis, had lower back pain that referred to the lower limbs, or those who had cardiovascular disease or other risk factor which precluded participation in aerobic exercise

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2020-01-18 (Actual); Study Completion 2020-01-18 (Actual)

PRIMARY OUTCOMES:
Change of quadriceps strength | Baseline and after six-week training
  Change from Baseline quadriceps strength after six-week training
Change of Functional questionnaire | Baseline and after six-week training
  Change from Baseline KOOS Chinese version after six-week training. The Knee Injury and Osteoarthritis Outcome Score (KOOS) is patient-administered that commonly used to evaluate the extent of knee pain and functional impairments in patients with different knee conditions, including knee OA. There are five subscales in this questionnaire.The score range is 0-100 and calculated for each subscale with lower score indicating extreme problems.
Change of Pain | Baseline and after six-week training
  Change from Baseline VAS scale after six-week training. A standard 10-centimeter visual analog scale (VAS) is a unidimensional measure of pain intensity. The score range is 0-10 with a higher score indicating greater pain intensity.

SECONDARY OUTCOMES:
Changes of thigh muscle activation | Baseline, after 3-week and six-week training
  Change from Baseline electromyography of vasti at 3-week and 6-week

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang CM, Chung H, Hsu HC, Chen LT, Lin RY, Lin HC. Effectiveness of stationary cycling with electromyographic biofeedback on neuromuscular control and function in individuals with knee osteoarthritis: a feasibility study. BMC Musculoskelet Disord. 2025 Jun 3;26(1):547. doi: 10.1186/s12891-025-08794-7. PMID 40462058